CLINICAL TRIAL: NCT05121922
Title: Sense of Coherence and Empowerment at Patients With Medically Unexplained Physical Symptoms in General Practice
Brief Title: Sense of Coherence and Empowerment at Patients With MUPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Erik L Werner, Professor, University of Oslo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IL001
Record Dates: First submitted 2021-10-19; First posted 2021-11-16 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Medically Unexplained Symptoms; Sense of Coherence
MeSH Terms: conditions — Medically Unexplained Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All patients recieve active treatment
  Interventions: Behavioral: Metacognitive Therapy

INTERVENTIONS:
Behavioral: Metacognitive Therapy — Psychological treatment provided by the patient's regular general practitioner

SUMMARY:
This is a study on Metacognitive therapy in general practice in Norway. The intervention is a small pilot study to examine whether Metacognitive therapy is feasible in an ordinary general practice. Will the physicians be capable to learn and provide the therapy method for their patients with MUPS and is is possible to implement this in an ordinary general practice routine? Both physicians and their patients will be asked to respond to a questionnaire on perceived utility of the treatment.

DETAILED DESCRIPTION:
Metacognitive therapy is different from Cognitive therapy in the sense that it adresses the individual's attention towards potential worries and threats and also the management performed by the patient to avoid these. Also the individual's capacity to produce empowerment to manage these threats are of interest in the talks with the health care provider. - In this study, General Practitioners with specific training in Metacognitive therapy will be asked to recruit 2-3 patients with Medically Unexplained Physical Symptoms each and invite them to a series of Metacognitive Therapy. The patients and physicians will then provide their assessments of the treatment on a number of questionnaires. To explore the Sense of coherence and Empowerment among patients with Medically Unexplained Symptoms, the physicians will be asked to recruit six patients each to respond to a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* MUPS: Medically Unexplained Physical Symptoms
* somatic and mental examination sufficiently accomplished
* ongoing symptoms
* more than three months of disabeling symptoms

Exclusion Criteria:

* not capable to respond on a written questionnaire in Norwegian

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility in daily practice | One year
  The physicians will record the number of patients that agree to participate and complete the treatment

SECONDARY OUTCOMES:
Effect of metacognitive therapy | One year
  Participating patients will respond on The Cognitive Attentional Syndrome Questionnaire (CAS-1) following each treatment session. A reduced score indicates improvement of symptom burden.
Effect of metacognitive therapy | One year
  Participating patients will respond on The Sense of Coherence Questionnaire (SOC-29) at start and at the end of the treatment. A reduced score indicates improvement of symptom burden.
Effect of metacognitive therapy | One year
  Participating patients will respond on The Short Form Health Survey RAND-36 at start and at the end of the treatment. A reduced score indicates improvement of symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Jørund Straand, PhD, Study Chair — University of Oslo
Locations (1):
- University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No